CLINICAL TRIAL: NCT03939234
Title: Peptide Vaccination With PD-L1 and PD-L2 Peptides in Untreated Chronic Lymphatic Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Møller Pedersen (Other)
Collaborators: IO Biotech (Industry)
Responsible Party: Sponsor-Investigator, Lars Møller Pedersen, Chief Phycisian, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL19H1; 2018-004869-14 (EudraCT Number)
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): Untreated CLL patients with unmutated IgHV gene with a cut of at maximum of 2 % mutations. According to guidelines from the European Research Initiative on CLL (ERIC).
  Interventions: Combination Product: PD-L1, PD-L2 peptides with Montanide ISA51

INTERVENTIONS:
Combination Product: PD-L1, PD-L2 peptides with Montanide ISA51 — PD-L1: 19 amino acid sequence from the PD-L1 protein; PD-L2: 21 amino acid sequence from the PD-L2 protein; The peptides are dissolved in dimethyl sulphoxide (DMSO) and mixed with Montanide.
  Other Names: IO103, IO120

SUMMARY:
This study is investigating the efficacy of PD-L1 and PD-L2 peptides in untreated CLL patients with unmutated IGHV gene status.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is an incurable disease with the unmutated immunoglobulin heavy chain variable region (IGHV) gene status being an unfavorable prognostic marker. These patients have shorter time to first treatment which consist of toxic chemotherapy.

Programmed death ligand 1 (PD-L1) and programmed death ligand 2 (PD-L2) are immune checkpoints hampering immune responses in many tumors including CLL. These proteins are expressed by suppressive bystander cells as well as CLL cells. Vaccinating subcutaneously with PD-L1 and PD-L2 peptides mobilises cytoxic T-cells specific towards PD-L1 and PD-L2 expressing cells. In this study we investigate if the PD-L1 and PD-L2 specific responses can overcome leukemic cells in CLL.

ELIGIBILITY:
Inclusion Criteria:

* CLL according to national guidelines (Lymphoma.dk).
* Unmutated IGHV gene according to ERIC recommendations.(25)
* No prior CLL directed treatment
* Age ≥ 18
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* No life-threatening conditions
* Adequate bone marrow function: Neutrophils > 1,0 x 109/l; Platelets > 100 x 109/l
* Adequate renal function: Glomeruli filtration rate (eGFR)/1,73 m2 > 50 mL/min
* Adequate liver function: Aspartate Aminotransferase < 100 U/L
* For fertile women: agreement to use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 120 days after the last treatment.
* For men: agreement to use contraceptive measures and agreement to refrain from donating sperm.

Exclusion Criteria:

* Other active malignant diseases requiring treatment.
* Significant medical condition per investigators judgement e.g. severe Asthma or chronic obstructive lung disease (COLD), poorly regulated heart condition, insulin dependent diabetes mellitus.
* Acute or chronic viral/bacterial infection e.g. human immunodeficiency virus (HIV), Cytomegalo virus (CMV), Epstein-barr virus (EBV), hepatitis or tuberculosis
* Serious known allergies or earlier anaphylactic reactions.
* Known sensibility towards Montanide ISA51
* Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
* Pregnant and breastfeeding women.
* Fertile women not using secure contraception with a failure rate less than < 1%
* Psychiatric disorders that according to the investigator could influence compliance.
* Treatment with other experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical response according to IW-CLL | 1 year
  Progressive disease (PD), stable disease (SD), partial response (PR), complete response (CR) calculated on basis of changes in circulating lymphocytes and lymphnode/spleen/liver size according to criteria from the international working group on CLL (IW-CLL).

SECONDARY OUTCOMES:
Immune response by elispot | 1 year
  T-cell responses measured by Enzyme-linked immunospot assay (ELISpot) counting the number of spots with cytokine release.
Grades of adverse events (AE) | 1 year
  Registered according to common terminology criteria for adverse events (CTCAE) v4.03. Each AE will be Graded I-V.

CONTACTS AND LOCATIONS:
Overall Officials: Uffe M Klausen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klausen U, Grauslund JH, Jorgensen NGD, Ahmad SM, Jonassen M, Weis-Banke SE, Martinenaite E, Pedersen LB, Lisle TL, Gang AO, Enggaard L, Hansen M, Holmstrom MO, Met O, Svane IM, Niemann CU, Pedersen LM, Andersen MH. Anti-PD-L1/PD-L2 therapeutic vaccination in untreated chronic lymphocytic leukemia patients with unmutated IgHV. Front Oncol. 2022 Nov 22;12:1023015. doi: 10.3389/fonc.2022.1023015. eCollection 2022. PMID 36483037